CLINICAL TRIAL: NCT00351013
Title: A Pilot Study of the Use of Homeopathic-Based Treatment Approaches to Reduce the Prevalence of Malaria in Depressed Communities
Brief Title: The Use of Homeopathic-Based Treatment Approaches to Reduce the Prevalence of Malaria in Depressed Communities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Malamed (Other)
Collaborators: Blackie Foundation Trust (Other)
Responsible Party: Dr. Jacob Minah, Malamed
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: BFT2006/2
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Malaria
Keywords: malaria; Plasmodium falciparum; Tropica Nosode; Homeopathy
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Malaria Tropica Nosode D200

INTERVENTIONS:
Other: Malaria Tropica Nosode D200 — 5 pellets every four months

SUMMARY:
Malaria accounts for over 40% of outpatient morbidity in Sierra Leone. These health risks have been heightened further by the recent civil war, persistent poverty, lack of access to affordable health care, and an increasing resistance of P.falciparum parasites to the most commonly used therapy Chloroquine, which now has a confirmed failure rate of 39%. This study will recruit 780 people from the Kroo-Bay community in Freetown. Healthy subjects would be randomised into two subgroups and given either homeopathic pellets or placebo tablets at four month intervals. They are then monitored repeatedly during the study period to assess the efficacy of the therapy in reducing the disease burden.

DETAILED DESCRIPTION:
The main objective of this project is to evaluate the efficacy, costs and benefits of homeopathic treatment therapies.This study will be conducted in the Kroo Bay community within Freetown, the capital city of Sierra Leone. This is a region where malaria is endemic with an annual average of one malaria episode per person.Further, given the high rates of poverty, most residents cannot afford to purchase the conventional drugs used to treat the malaria. Chloroquine, which is the cheapest drug available, is no longer efficacious for P.falciparum parasites.

The study will utilize a longitudinal approach that is divided into three major phases. The first is a pre-test period involving the preparation and review of protocols, staff training, purchase of equipment and medical supplies. Phase two constitutes an open randomised controlled trial phase that is divided into five stages. The first stage IIA involves subject recruitment from the Kroo-Bay community in the capital city of Freetown. Approximately 780 permanent residents (ages 18+) living within a radius of 10 km within the community would be recruited. A questionnaire would be administered to evaluate personal case histories, use of mosquito bed nets, frequency of malaria diagnoses, the kinds of treatments used in the past, and knowledge of alternative treatment therapies. Other variables such as age, height, weight, gender, occupation and socio-economic attributes would be collected. All subjects would be tested for malaria using blood smears. Those who test positive for malaria, with clinical symptoms such as high temperature (>37.5 C) and high levels of parasitemia (asexual forms of P falciparum >5000ul blood) would be sent to the local clinic for treatment. These individuals would constitute the first subgroup in the study sample. The remaining subjects eligible for the clinical trial would be those with no major underlying illnesses, normal body temperatures and a reduced load of asexual forms of P falciparum < 5000ul blood). All subjects would be monitored for four months and asked to return for their second prophylactic treatment in four months (Day 112).

The next stage (IIB) begins after four months during which subjects are retested for malaria and based on their blood sample results (negative), healthy subjects would be given another dose of the pellets. They will be monitored for another four months. The same protocol is followed in the next three consecutive stages (IIC, IID, and IIE). During each follow-up visit, the subjects are retested and those with negative results are placed on their regimen for four months.

The clinical trial phase ends after stage IIE. In the third phase, a post-intervention survey will be given to all subjects to evaluate the levels of awareness of malaria and knowledge of alternative treatment remedies. All data measures including, residential location, blood test results, health histories and socio-demographic attributes would be compiled and analyzed statistically to evaluate the effectiveness of the homeopathic treatment. The results are expected to be published in a scientific peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate:
* Ability to understand and sign consent form,
* Permanent residence within 10km radius of Kroo Bay

Exclusion Criteria:

* Serious Underlying Illness,
* Absence from the study for 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2006-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
reduction in the burden and severity of malaria episodes | four months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Minah, MD, Principal Investigator — Specialist Pediatrician, Homeopath, Germany; Florence M. Margai, PhD, Principal Investigator — Professor, Binghamton University-New York
Locations (1):
- Malamed, Freetown, Sierra Leone